CLINICAL TRIAL: NCT00517634
Title: A 12-week, Randomised, Double-blind, Placebo-controlled, Three-period, Cross-over Pilot Study Comparing the Effect of Salmeterol/Fluticasone Propionate, Fluticasone Propionate and Placebo on Perpheral Blood Eosinophils and Serum IL-5 in Response to Allergen Challenge in Asthma Subjects When Allergen Challenge is Administered at 1 Hour or 11-12 Hours Post-dose of the Dosing Interval
Brief Title: Study Of Fluticasone Propionate/Salmeterol In Asthmatic Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HZA109912
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Results first posted 2009-09-02 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: asthma; allergen challenge; IL-5; eosinophils
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1: FP, SFC, Placebo (Experimental): Fluticasone Propionate (FP) 100 micrograms (mcg) twice daily (BID) in the first treatment period: Salmeterol/Fluticasone Propionate Combination (SFC) 50/100 mcg BID in the second treatment period: Placebo in the third treatment period
  Interventions: Drug: FP; Drug: SFC; Drug: Placebo
- Sequence 2: Placebo, SFC, FP (Experimental): Placebo in the first treatment period: Salmeterol/Fluticasone Propionate Combination 50/100 mcg BID in the second treatment period: Fluticasone Propionate 100 mcg BID in the third treatment period
  Interventions: Drug: FP; Drug: SFC; Drug: Placebo
- Sequence 3: SFC, FP, Placebo (Experimental): Salmeterol/Fluticasone Propionate 50/100 Combination mcg BID in the first treatment period: Fluticasone Propionate 100 mcg BID in the second treatment period: Placebo in the third treatment period
  Interventions: Drug: FP; Drug: SFC; Drug: Placebo
- Sequence 4: SFC, Placebo, FP (Experimental): Salmeterol/Fluticasone Propionate Combination 50/100 mcg BID in the first treatment period: Placebo in the second treatment period: Fluticasone Propionate 100 mcg BID in the third treatment period
  Interventions: Drug: FP; Drug: SFC; Drug: Placebo
- Sequence 5: FP, Placebo, SFC (Experimental): Fluticasone Propionate 100 mcg BID in the first treatment period: Placebo in the second treatment period: Salmeterol/Fluticasone Propionate Combination 50/100 mcg BID in the third treatment period
  Interventions: Drug: FP; Drug: SFC; Drug: Placebo
- Sequence 6: Placebo, FP, SFC (Experimental): Placebo in the first treatment period: Fluticasone Propionate 100 mcg BID in the second treatment period: Salmeterol/Fluticasone Propionate Combination 50/100 mcg BID in the third treatment period
  Interventions: Drug: FP; Drug: SFC; Drug: Placebo

INTERVENTIONS:
Drug: FP — Fluticasone Propionate 100 mcg BD
Drug: SFC — Salmeterol/Fluticasone Propionate Combination 50/100 mcg BD
Drug: Placebo — Matching Placebo

SUMMARY:
The aim of the present study is to investigate whether the effects of salmeterol in combination with fluticasone propionate on blood markers of airway inflammation are maintained after chronic dosing and whether the effect is influenced by the time of allergen challenge relative to the time of dosing.

DETAILED DESCRIPTION:
A 12-week, randomised, double-blind, placebo-controlled, three-period, cross-over pilot study comparing the effect of salmeterol/fluticasone propionate, fluticasone propionate and placebo on perpheral blood eosinophils and serum IL-5 in response to allergen challenge in asthma subjects when allergen challenge is administered at 1 hour or 11-12 hours post-dose of the dosing interval

ELIGIBILITY:
Inclusion Criteria:

* Informed consent.
* Outpatient.
* Male or non-pregnant/non-lactating female.
* Aged 18-55.
* Diagnosis of asthma.
* Pre-bronchodilatory FEV1 > 75% predicted.
* Using inhaled short-acting beta-2-agonists (SABA) with no inhaled corticosteroids.
* Judged capable of withholding SABA for at least 6 hours prior to visits.
* Reversibility of >12% and 200mL or PC20 of <8mg/mL.
* Demonstration of atopy

Exclusion Criteria:

* History of life-threatening asthma.
* Use of proscribed asthma medications.
* Use of anti-histamines or potent inhibitors of CYP3A4.
* Respiratory tract infection.
* Asthma exacerbation with 4 weeks of Visit 1.
* Subjects with exercise induced asthma only.
* Concurrent respiratory disease.
* Other clinically significant, uncontrolled condition or disease.
* Use of any investigational drug within 30 days.
* Allergic to beta-2-agonists, inhaled corticosteroids or excipients.
* Positive pregnancy test.
* Using immunosuppressive medications.
* Milk protein allergy.
* Factors likely to interfere with attendance.
* Current smokers or ex-smokers with a history of >10 pack years.
* Affiliation wih Investigator site.
* Medications that may affect the course of asthma or interact with sympathomimetic amines.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Madison, Wisconsin, United States
- GSK Investigational Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: HZA109912 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: HZA109912 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: HZA109912 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: HZA109912 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: HZA109912 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: HZA109912 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: HZA109912 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: First Treatment Period
Arm/Group | Sequence 1: FP, SFC, Placebo | Sequence 2: Placebo, SFC, FP | Sequence 3: SFC, FP, Placebo | Sequence 4: SFC, Placebo, FP | Sequence 5: FP, Placebo, SFC | Sequence 6: Placebo, FP, SFC
Started | 4 | 4 | 4 | 3 | 4 | 4
Completed | 4 | 4 | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Treatment Period
Arm/Group | Sequence 1: FP, SFC, Placebo | Sequence 2: Placebo, SFC, FP | Sequence 3: SFC, FP, Placebo | Sequence 4: SFC, Placebo, FP | Sequence 5: FP, Placebo, SFC | Sequence 6: Placebo, FP, SFC
Started | 4 | 4 | 4 | 3 | 4 | 4
Completed | 4 | 4 | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Third Treatment Period
Arm/Group | Sequence 1: FP, SFC, Placebo | Sequence 2: Placebo, SFC, FP | Sequence 3: SFC, FP, Placebo | Sequence 4: SFC, Placebo, FP | Sequence 5: FP, Placebo, SFC | Sequence 6: Placebo, FP, SFC
Started | 4 | 4 | 4 | 3 | 3 | 4
Completed | 4 | 4 | 4 | 3 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: Overall Study Population: participants in all three treatment periods
Arm/Group | Overall Study Population
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (6.63)
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 14
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 2
  Caucasian | 21

OUTCOME MEASURES:

1. Primary Outcome: Weighted Mean Change From Baseline Over 0-6 Hours in Blood Eosinophils Post-Allergen Challenge on Day 35
Description: Number of peripheral blood eosinophils measured from blood draws
Time Frame: 0-6 hours post allergen challenge, 10-11 hours post treatment, Day 35
Population: Intent-to-Treat (ITT) Population: All participants receiving at least one dose of study medication who had at least one post-randomization efficacy assessment
Measure: Mean (95% Confidence Interval); unit: Giga Units per Liter (GI/L)
Groups:
- Placebo: Placebo
- FP 100 mcg BID: Fluticasone Propionate (FP) 100 mcg BID
- SFC 50/100 mcg BID: Salmeterol/Fluticasone Propionate Combination (SFC) 50/100 mcg BID
Arm/Group | Placebo | FP 100 mcg BID | SFC 50/100 mcg BID
Number analyzed (Participants) | 22 | 22 | 22
Giga Units per Liter (GI/L) | -0.050 [-0.072 to -0.029] | -0.040 [-0.061 to -0.019] | -0.023 [-0.044 to -0.001]

2. Secondary Outcome: Weighted Mean Change From Baseline Over 0-6 Hours in Blood Eosinophils Post-Allergen Challenge on Day 14
Description: Number of peripheral blood eosinophils measured from blood draws
Time Frame: 0-6 hours, post allergen challenge, 1 hour post treatment, Day 14
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: Giga Units per Liter (GI/L)
Arm/Group | Placebo | FP 100 mcg BID | SFC 50/100 mcg BID
Number analyzed (Participants) | 21 | 23 | 20
Giga Units per Liter (GI/L) | -0.023 [-0.039 to -0.006] | -0.022 [-0.038 to -0.007] | -0.013 [-0.029 to -0.004]

3. Secondary Outcome: Weighted Mean Change From Baseline Over 0-6 Hours in Serum IL-5 Post-Allergen Challenge on Day 35
Description: Amount of serum interleukin (IL)-5 measured from blood draws
Time Frame: 0-6 hours post allergen challenge, 10-11 hours post treatment, Day 35
Reporting Status: Not Posted

4. Secondary Outcome: Weighted Mean Change From Baseline Over 0-6 Hours in Serum IL-5 Post-Allergen Challenge on Day 14
Description: Amount of serum IL-5 measured from blood draws
Time Frame: 0-6 hours post allergen challenge, 1 hour after dosing, Day 14
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- FP 100 mcg BID: Fluticasone Propionate 100 mcg BID
- SFC 50/100 BID: Salmeterol/Fluticasone Propionate Combination 50/100 mcg BID
Arm/Group | Placebo | FP 100 mcg BID | SFC 50/100 BID
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 1/22
Other Adverse Events (participants affected / at risk) | 14/22 | 16/23 | 10/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | FP 100 mcg BID (N=23) | SFC 50/100 BID (N=22)
Appendicitis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | FP 100 mcg BID (N=23) | SFC 50/100 BID (N=22)
Headache (Nervous system disorders) | 7 | 3 | 2
Nasopharyngitis (Infections and infestations) | 2 | 3 | 2
Pharyngolarngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0
Discomfort (General disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Multiple allergies (Immune system disorders) | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
House dust allergy (Immune system disorders) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.